CLINICAL TRIAL: NCT01293448
Title: Evaluation of Balloon-based Cryoablation of Human Esophageal Epithelium
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pentax Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-0001.A
Record Dates: First submitted 2010-12-14; First posted 2011-02-10 (Estimated); Last update posted 2022-04-28 (Actual); Status verified 2018-01

CONDITIONS: Barrett's Esophagus; Esophageal Cancer
Keywords: Esophagectomy; Barrett's Esophagus
MeSH Terms: conditions — Barrett Esophagus; Esophageal Neoplasms | interventions — Cryosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): CryoBalloon ablation of esophageal tissue in patients scheduled for esophagectomy for reasons unrelated to the objective of the study.
  Interventions: Device: Cryoballoon Ablation

INTERVENTIONS:
Device: Cryoballoon Ablation — Device: CryoBalloon Ablation System(TM) C2 Therapeutics Inc. received FDA market clearance for the CryoBalloon Ablation System on September 29, 2010. The System is a Class II device "intended to be used as a cryosurgical tool for the destruction of unwanted tissue in the field of general surgery, specifically for endoscopic applications." (K101825)
  Other Names: CryoBalloon Ablation System; cryoablation

SUMMARY:
The purpose of this study is to evaluate a cryoablation technique used to ablate human esophageal mucosa.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the histological results of a cryoablation technique used to ablate human esophageal mucosa. The performance and safety of the cryoablation technique will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have a minimum of 2.0 cm of non-ulcerated, non-inflammatory columnar-lined esophagus or squamous esophageal lined tissue suitable for ablation. A patient may be treated with up to 2 zones of ablation.
* Patient is 18 to 80 years of age at the time of consent (inclusive).
* Patient has provided written Informed Consent Form (IFC) using a form that has been approved by the Institution's reviewing IRB/EC.
* Patient is willing and able to comply with all Clinical Investigation Plan (CIP) requirements.
* Patient's esophagectomy is clinically necessary due to reasons unrelated to this study.
* Patient is deemed operable per standard institutional criteria.

Exclusion Criteria:

* Patient has a known history of unresolved drug or alcohol dependency that would limit ability to comprehend or follow instructions related to IFC, post treatment instructions or follow-up guidelines.
* Patient refuses or is unable to provide written informed consent. - -
* Patient has or is currently undergoing endoscopic ablation therapy within 4 cm from the proposed treatment area including, but not limited to cryospray therapy, laser treatment, photodynamic therapy, multi-polar electro coagulation, endoscopic mucosal resection, radiofrequency ablation or argon plasma coagulation.
* Patient has esophageal narrowing limiting access to the intended site of ablation.
* Patient is undergoing or has recently undergone chemotherapy (within 15 days or WBC below normal by institutional criteria or standards).
* Patient is undergoing or has recently undergone radiation therapy which involved the esophagus (within 15 days or WBC below normal by institutional criteria or standards).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-12; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Treatment effect | Within 30 days of ablation procedure
  The primary outcome measure is to evaluate the histological results (depth of injury) of a cryoballoon ablation system.

SECONDARY OUTCOMES:
Post-ablation symptoms | Within 7 days of ablation procedure
  A secondary outcome measure is to evaluate post-ablation symptoms - number of participants with adverse events as a measure of safety and tolerability.
Post procedure pain | Within 7 days of ablation procedure
  The secondary objective of the study is to determine patient comfort post-procedure. Pain scores are measured on a numerical pain intensity scale.

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Bergman, MD, Principal Investigator — AIDS Malignancy Consortium; Steve DeMeester, MD, Principal Investigator — University of Southern California; Blair Jobe, MD, Principal Investigator — University of Pittsburgh; Jeffery Peters, MD, Principal Investigator — University of Rochester
Locations (4):
- United States (3):
  - University of Southern California, Los Angeles, California
  - University of Rochester, Rochester, New York
  - University of Pittsburgh, Pittsburgh, Pennsylvania
- AMC, Amsterdam, AZ, Netherlands